CLINICAL TRIAL: NCT06166355
Title: Improving the Treatment of Anorexia Nervosa in Children Through Virtual Reality Body Exposure
Acronym: EOAN-VR-ABM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Barcelona (Other)
Collaborators: Hospital Sant Joan de Deu (Other)
Responsible Party: Principal Investigator, Jose Gutierrez Maldonado, Professor, University of Barcelona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 510/U/2022
Record Dates: First submitted 2023-12-04; First posted 2023-12-12 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Anorexia Nervosa
Keywords: Attentional Bias; Virtual Reality; Eye-Tracking; Body exposure procedure; Attentional bias modification training
MeSH Terms: conditions — Anorexia Nervosa | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cognitive-behavioral therapy plus VR-based body exposure and Attentional Bias Modification Training. (Experimental): In this group, five sessions of VRE will be added to the usual CBT, as in the other experimental group, but, in addition, at the beginning of each of the exposure sessions, the training aimed at reducing the attentional bias will be carried out. The training will be developed through the visual selection of geometric figures that fit approximately with specific parts of the body. Each of these figures can have different colors. Specifically, the patient must detect and identify the figures that will appear in different parts of the avatar's body. In half of the trials, the shape of the figure must be discriminated and in the remaining 50%, the discrimination will be based on color. Throughout the training, the geometric figures will appear on weight-related body parts in 45% of the trials, and in another 45% of the trials, it will appear on non-weight-related body parts. In the remaining trials (10%), the test will appear on one of three neutral stimuli located next to the avatar.
  Interventions: Behavioral: Attentional Bias Modification Training; Behavioral: VR-based body exposure; Behavioral: Cognitive-behavioral therapy
- Cognitive-behavioral therapy for anorexia and VR-based body exposure: (Experimental): Patients assigned to this group will receive the usual CBT from the clinical unit or the hospital where they are, and additionally, five sessions of VR-based body exposure intervention. In these weekly sessions patients will go through a body exposure intervention in which they will own a virtual avatar with their real measurements, that will progressively increase its BMI values throughout the following exposure sessions until a healthy BMI value is reached.
  Interventions: Behavioral: VR-based body exposure; Behavioral: Cognitive-behavioral therapy
- Cognitive behavioral therapy (Active Comparator): Patients assigned to this group will receive the usual treatment from the center in which they are recruited for the study (CBT), and will have to complete the evaluations following the same schedule as the experimental group.
  Interventions: Behavioral: Cognitive-behavioral therapy

INTERVENTIONS:
Behavioral: Attentional Bias Modification Training — Combine usual cognitive-behavioral treatment (CBT) sessions with additional five VR-based body-exposure therapy sessions and five sessions of Attentional Bias Modification Training.
  Arms: Cognitive-behavioral therapy plus VR-based body exposure and Attentional Bias Modification Training.
Behavioral: VR-based body exposure — Combine usual cognitive-behavioral treatment (CBT) sessions with additional five VR-based body-exposure therapy sessions
  Arms: Cognitive-behavioral therapy for anorexia and VR-based body exposure:; Cognitive-behavioral therapy plus VR-based body exposure and Attentional Bias Modification Training.
Behavioral: Cognitive-behavioral therapy — Usual cognitive-behavioral treatment (CBT) sessions.

SUMMARY:
The age of onset of anorexia nervosa has been progressively decreasing in recent years. Also, the prevalence rates of childhood anorexia in many countries have grown significantly. This increase was already observed before the COVID-19 pandemic, but the confinements and the stress derived from them have caused this increase to accelerate. As in adolescent and adult patients, in childhood anorexia some of the core signs and symptoms are an extreme fear of gaining weight and avoidance of food. The consequences of the early-onset of anorexia can be very important since the maturation of the organism is more incomplete in children than in adolescents. Weight loss can have very severe consequences, since in children the percentage of body fat is lower. On the other hand, hormonal disorders derived from food deprivation also have very severe consequences for the development of different organs. General physical development and growth can be affected, with consequences such as not being able to reach normal height. The research carried out to date on the efficacy of treatments for childhood anorexia is very scarce. There are no specific treatment strategies or settings for children with anorexia, and little research has been done to tailor treatment for younger patients. Given the need to explore new treatments for anorexia nervosa specifically aimed at children, the objective of this project is to develop a program to carry out exposure to one's own body through virtual reality, gradually, with progressive increases in size until achieving a healthy weight. In the virtual exposure, patients will observe the image of an avatar in a mirror for the time necessary in each session to produce the reduction of the anxiety response. The avatars that will be developed for this purpose will have a physical constitution corresponding to children under 14 years of age, and physical proportions equivalent to those of each patient. The positive results obtained with a previous version of this treatment originally developed for adolescents and adults suggest that its adaptation to children can open new ways for exploring effective treatments for childhood anorexia.

DETAILED DESCRIPTION:
The age of onset of anorexia nervosa (AN) has been progressively decreasing in recent years, and the prevalence of childhood AN has grown significantly. This increase was already observed before the COVID-19 pandemic, but the confinements have caused this increase to accelerate. The incidence of eating disorders (ED) was 15.3% higher in 2020 compared with previous years. The relative risk increased steadily from March 2020 onwards, exceeding 1.5 by the end of the year. The increase was primarily related to teenagers and AN. A higher proportion of patients in 2020 had suicidal ideation or attempted suicide. Although the diagnostic criteria of AN are applied equally regardless of age, there are differential characteristics between child patients and adolescents or adults in the form of presentation, epidemiology, comorbidity and, also, in outcomes. In most studies, an age of less than 14 has been used as a criterion to define the childhood presentation of this disorder, since it coincides with the legal criterion in many countries. The somatic and mental consequences of early-onset anorexia have a strong negative effect on later adult life. Regardless of the treatment applied, only about half of patients maintain their restored weight in the long term. Little research has been done to tailor treatment for younger patients. Therefore, there is an urgent need for studies on new strategies to treat this serious disorder in children. The objective of this project is to develop a program to carry out exposure to one's own body through virtual reality, with progressive increases in the body mass index (BMI). Patients will observe an avatar in a mirror for the time necessary in each session to produce habituation, extinguishing the anxiety response. The avatars will have a physical constitution corresponding to children under 14 years old, and physical proportions equivalent to those of each patient. The results obtained with the version of this treatment originally developed for adolescents and adults by the investigation group suggest that its adaptation to children can open new ways for exploring effective treatments for children AN. It will also be analyzed whether the addition of a component aimed at modifying attentional biases towards the body increases the efficacy of the exposure. The hypothesis is: if a component of virtual-reality body exposure is added to the usual treatment for AN in children, then the treatment will be more effective. Furthermore, if a component designed to reduce body attention bias is also added, then the efficacy of the treatment will be even greater. The efficacy of this treatment, aimed at reducing the fear of gaining weight, will be analyzed in a randomized controlled study in which a group of patients under 14 years of age will receive treatment as usual, another group will receive treatment as usual plus five booster sessions of virtual body exposure, and a third group will receive treatment as usual, plus five booster sessions of virtual body exposure plus modification of attentional biases towards the body.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a primary diagnosis of anorexia nervosa (DSM-V)
* Patients below 14 years old
* Patients with BMI <18.5
* Subsyndromal patients will also be included

Exclusion Criteria:

* Visual deficits
* Epilepsy or neuroleptic medication
* Psychotic disorder
* Bipolar disorder
* Medical complications
* Pregnancy
* Clinical cardiac arrhythmia

Max Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 108 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Change in Eating Disorder symptomatology: Eating Disorders Inventory-3 (EDI-3; Garner, 2004) drive for thinness (EDI-DT) scale | From pre-assessment to post-assessment after 6 weeks , and at the six-month follow-up
  Evaluation of the change in drive for thinness, with maximum possible score of 28, where higher scores indicate higher drive for thinness.
Change in Eating Disorder symptomatology: Eating Disorders Inventory-3 (EDI-3; Garner, 2004) body dissatisfaction (EDI-BD) scale | From pre-assessment to post-assessment after 6 weeks , and at the six-month follow-up
  Evaluation of the change in body dissatisfaction, with maximum possible score of 40, where higher scores indicate higher body dissatisfaction.
Change in body mass index values | From pre-assessment to post-assessment after 6 weeks , and at the six-month follow-up
  Evaluation of change in Body Mass Index values

SECONDARY OUTCOMES:
Change in Body Anxiety: Physical Appearance State Anxiety Scale (PASTAS) | From pre-assessment to post-assessment after 6 weeks , and at the six-month follow-up
  Evaluation of body-related anxiety using the PASTAS, with a maximum score of 32, with higher scores indicating higher body-related anxiety
Change in Body image disturbance: Body Appreciation Scale (BAS) | From pre-assessment to post-assessment after 6 weeks , and at the six-month follow-up
  Evaluation of the change in body appreciation using the BAS, with a scale of possible scores ranging from 13-65, where higher scores indicate higher body appreciation
Change in Body image disturbance: Figural Drawing Scale for Body Image Assessment (BIAS-BD) body distortion scores | From pre-assessment to post-assessment after 6 weeks , and at the six-month follow-up
  Evaluation of the change in body distortion using the BIAS-BD body distortion scores, ranging from -80 to 80, with higher scores indicating higher body distortion
Change in Body image disturbance: Figural Drawing Scale for Body Image Assessment (BIAS-BD) body dissatisfaction scores | From pre-assessment to post-assessment after 6 weeks , and at the six-month follow-up
  Evaluation of the change in body dissatisfaction using the BIAS-BD body dissatisfaction scores, ranging from -80 to 80, with higher scores indicating higher body dissatisfaction
Change in complete fixation time of the gaze towards weight-related body parts | From pre-assessment to post-assessment after 6 weeks
  Evaluation of the attentional bias towards the body using complete fixation time (evaluated in milliseconds) of the gaze towards weight-related body parts, with higher values indicating a greater attentional bias.
Change in number of fixations of the gaze towards weight-related body parts | From pre-assessment to post-assessment after 6 weeks
  Evaluation of the attentional bias towards the body using number of fixations of the gaze towards weight-related body parts, with higher values indicating a greater attentional bias

OTHER OUTCOMES:
Body-related anxiety | Up to 40 minutes. Baseline (prior to beginning the body exposure session), every two minutes during the exposure, and at the end of the body exposure session
  Visual analogue scale from 0 to 100, with higher scores indicating higher body-related anxiety
Fear of gaining weight | Up to 40 minutes. Baseline (prior to beginning the body exposure session) and at the end of the body exposure session
  Visual analogue scale from 0 to 100, with higher scores indicating higher fear of gaining weight
Full body ownership illusion | Up to 40 minutes. Baseline (prior to beginning the body exposure session) and at the end of the body exposure session
  Visual analogue scale from 0 to 100, with higher scores indicating higher full body ownership illusion

CONTACTS AND LOCATIONS:
Overall Officials: José Gutiérrez-Maldonado, Principal Investigator — University of Barcelona
Locations (1):
- Hospital Sant Joan de Déu, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
The data presented in this study will be available on request from the corresponding author. The data are not publicly available due to patients' privacy restrictions.